CLINICAL TRIAL: NCT02630706
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, 26-Week Multicenter Study to Evaluate the Efficacy and Safety of Ertugliflozin in Asian Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control on Metformin Monotherapy (VERTIS-ASIA)
Brief Title: A Study to Evaluate the Efficacy and Safety of Ertugliflozin in Asian Participants With Type 2 Diabetes and Inadequate Glycemic Control on Metformin Monotherapy (MK-8835-012)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8835-012; B1521045 (Other: Pfizer Protocol Number); MK-8835-012 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Results first posted 2018-12-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ertugliflozin; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor was masked.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ertugliflozin 5 mg (Experimental): Ertugliflozin 5 mg oral and matching placebo for ertugliflozin 10 mg, oral, once daily for 26 weeks, while maintaining metformin at a stable dose (>=1500 mg/day). Glycemic rescue therapy with open-label glimepiride was initiated in participants with glucose values exceeding protocol-specified values.
  Interventions: Drug: Ertugliflozin 5 mg; Drug: Placebo matching ertugliflozin; Drug: Metformin; Drug: Glimepiride
- Ertugliflozin 15 mg (Experimental): Ertugliflozin 15 mg (ertugliflozin 5 mg + ertugliflozin 10 mg) administered orally once daily for 26 weeks, while maintaining metformin at a stable dose (>=1500 mg/day). Glycemic rescue therapy with open-label glimepiride was initiated in participants with glucose values exceeding protocol-specified values.
  Interventions: Drug: Ertugliflozin 15 mg; Drug: Metformin; Drug: Glimepiride
- Placebo (Placebo Comparator): Placebo matching ertugliflozin administered orally once daily for 26 weeks, while maintaining metformin at a stable dose (>=1500 mg/day). Glycemic rescue therapy with open-label glimepiride was initiated in participants with glucose values exceeding protocol-specified values.
  Interventions: Drug: Placebo matching ertugliflozin; Drug: Metformin; Drug: Glimepiride

INTERVENTIONS:
Drug: Ertugliflozin 5 mg — Ertugliflozin 5 mg oral tablet taken once daily
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 5 mg
Drug: Ertugliflozin 15 mg — Ertugliflozin 15 mg (5-mg and 10-mg tablets) oral taken once daily
  Other Names: MK-8835; PF-04971729
  Arms: Ertugliflozin 15 mg
Drug: Placebo matching ertugliflozin — Placebo matching ertugliflozin (5-mg and/or 10-mg tablet) oral taken once daily
  Arms: Ertugliflozin 5 mg; Placebo
Drug: Metformin — Participants are to remain on their stable doses of metformin (oral, >=1500 mg/day) while receiving blinded investigational product during the double-blind treatment period. Participants on metformin <1500 at screening are up-titrated to >= 1500 daily.
Drug: Glimepiride — Glycemic rescue therapy with open-label glimepiride will be initiated in participants with glucose values exceeding protocol-specified values. Dosing and titration of open-label glimepiride rescue therapy will be at the Investigator's discretion.

SUMMARY:
This is a study to evaluate the efficacy and safety of the addition of ertugliflozin to metformin monotherapy in Asian participants with Type 2 diabetes mellitis (T2DM) who have inadequate glycemic control on metformin monotherapy. The primary hypothesis is that the mean reduction from baseline in HbA1C for 15 mg and 5 mg ertugliflozin (tested sequentially) is greater than for placebo.

DETAILED DESCRIPTION:
This study includes a 1-week screening period, an 8-week (or greater) antihyperglycemic agent (AHA) wash-off and/or metformin dose stable period (as necessary), a 2-week single-blind placebo run-in period, a 26-week double-blind treatment period, and a post-treatment telephone contact 14 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Asian participants ≥18 years of age at the time of initial Screening.
* Type 2 diabetes mellitus as per American Diabetes Association guidelines.
* Metformin monotherapy (≥1500 mg/day) with an initial Screening A1C of 7.0-10.5% (53-91 mmol/mol) OR metformin monotherapy (<1500 mg/day) with an initial Screening A1C of 7.5-11.0% (58-97 mmol/mol) OR dual combination therapy with metformin + sulfonylurea, dipeptidyl peptidase-4 (DDP-4) inhibitor, meglitinide, or alpha-glucosidase inhibitor with an initial Screening A1C of 6.5-9.5% (48-80 mmol/mol).
* Body mass index (BMI) ≥18.0 kg/m^2.
* Male or female not of reproductive potential.
* Female of reproductive potential who agrees to remain abstinent from heterosexual activity or to use 2 acceptable combinations of contraception.

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis.
* History of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post-organ transplant.)
* History of myocardial infarction, unstable angina, arterial revascularization, stroke, transient ischemic attack, or New York Heart Association (NYHA) functional class III-IV heart failure within 3 months of study start.
* Mean value for triplicate screening sitting systolic blood pressure >160 mm Hg and/or diastolic blood pressure >90 mm Hg after at least a 5-minute seated rest at screening
* Active, obstructive uropathy or indwelling urinary catheter.
* History of malignancy ≤5 years prior to study start, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week or engages in binge drinking.
* Any clinically significant malabsorption condition.
* Is on a weight-loss program or weight-loss medication or other medication associated with weight changes and is not weight stable prior to study start.
* Has undergone bariatric surgery within the past 12 months or >12 months and is not weight stable prior to study start.
* A known hypersensitivity or intolerance to any sodium glucose co-transporter (SGLT2) inhibitor.
* On a previous clinical study with ertugliflozin.
* Is taking blood pressure or lipid altering medications that have not been on a stable dose for at least 4 weeks prior to study start.
* Current treatment for hyperthyroidism.
* Male participants with a serum creatinine >=1.3 mg/dL (>=115 mol/L) or female participants with a serum creatinine >=1.2 mg/dL (>=106 mol/L) or participants with an estimated glomerular filtration rate (eGFR) <55 mL/min/1.73m^2 according to the 4-variable Modification of Diet in Renal Disease (MDRD) equation at screening.
* An aspartate transaminase (AST) or alanine transaminase (ALT) >2X the upper limit of normal (ULN) range at screening, or a total bilirubin >1.5 X the ULN unless the participant has a history of Gilbert's.
* On thyroid replacement therapy and has not been on a stable dose for at least 6 weeks prior to study start.
* A medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease.
* Has been treated with any of the following agents within 12 weeks of study start or during the pre-randomization period: Insulin of any type (except for short-term use during concomitant illness or other stress), other injectable anti-hyperglycemic agents (e.g., pramlintide, exenatide, liraglutide), another SGLT2 inhibitor, bromocriptine, colesevelam, rosiglitazone or pioglitazone, or any other AHA with the exception of the protocol-approved agents.
* Is on or likely to require treatment ≥14 consecutive days or repeated courses of pharmacologic doses of corticosteroids.
* Has undergone a surgical procedure within 6 weeks prior to study start or has planned major surgery during the study.
* Pregnant or breast-feeding, or planning to conceive during the trial, including 14 days following the last dose of study medication.
* Planning to undergo hormonal therapy in preparation for egg donation during the trial, including 14 days following the last dose of study medication.
* Donated blood or blood products within 6 weeks of study start.
* Has Human Immunodeficiency Virus (HIV).
* Has blood dyscrasias or any disorders causing hemolysis or unstable red blood cells.
* Has clinically important hematological disorders (such as aplastic anemia, myeloproliferative or myelodyplastic syndromes, thrombocytopenia.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ji L, Liu J, Xu ZJ, Wei Z, Zhang R, Malkani S, Cater NB, Frederich R. Efficacy and Safety of Ertugliflozin Added to Metformin: A Pooled Population from Asia with Type 2 Diabetes and Overweight or Obesity. Diabetes Ther. 2023 Feb;14(2):319-334. doi: 10.1007/s13300-022-01345-6. Epub 2023 Feb 3. PMID 36763328
- [Derived] Xu H, O'Gorman MT, Nepal S, James LP, Ginman K, Pithavala YK. Phase 1 Study Evaluating the Effects of the Proton Pump Inhibitor Rabeprazole and Food on the Pharmacokinetics of Lorlatinib in Healthy Participants. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1395-1404. doi: 10.1002/cpdd.1000. Epub 2021 Jul 20. PMID 34288547
- [Derived] Fediuk DJ, Sahasrabudhe V, Dawra VK, Zhou S, Sweeney K. Population Pharmacokinetic Analyses of Ertugliflozin in Select Ethnic Populations. Clin Pharmacol Drug Dev. 2021 Nov;10(11):1297-1306. doi: 10.1002/cpdd.970. Epub 2021 Jul 2. PMID 34213819
- [Derived] Ji L, Liu Y, Miao H, Xie Y, Yang M, Wang W, Mu Y, Yan P, Pan S, Lauring B, Liu S, Huyck S, Qiu Y, Terra SG. Safety and efficacy of ertugliflozin in Asian patients with type 2 diabetes mellitus inadequately controlled with metformin monotherapy: VERTIS Asia. Diabetes Obes Metab. 2019 Jun;21(6):1474-1482. doi: 10.1111/dom.13681. Epub 2019 Apr 5. PMID 30830724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 1078 participants were screened, and 506 participants were randomized at 50 sites in China, Hong Kong, Republic of Korea, the Philippines, and Taiwan.
Groups:
- Ertugliflozin 15 mg: Ertugliflozin 15 mg administered orally once daily for 26 weeks, while maintaining metformin at a stable dose (>=1500 mg/day). Glycemic rescue therapy with open-label glimepiride was initiated in participants with glucose values exceeding protocol-specified values.
Period: Overall Study
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Started | 170 | 169 | 167
Treated | 170 | 169 | 167
Completed | 163 | 160 | 157
Not Completed | 7 | 9 | 10
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 7

BASELINE CHARACTERISTICS:
Population: The analysis population included all randomized participants who received at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo | Total
Number analyzed (Participants) | 170 | 169 | 167 | 506
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (9.0) | 56.3 (9.3) | 56.9 (9.0) | 56.5 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  Participants
    Female | 75 | 71 | 79 | 225
    Male | 95 | 98 | 88 | 281
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 170 | 169 | 167 | 506
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  Kilograms | 71.4 (11.1) | 69.5 (10.9) | 70.1 (12.4) | 70.3 (11.5)
Baseline Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percentage A1C] — Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Population: The analysis population included all randomized participants who have received at least one dose of investigational product and had a baseline A1C measurement.
  Percentage A1C
    number analyzed (Participants) | 169 | 169 | 166 | 504
    (all) | 8.14 (0.89) | 8.09 (0.91) | 8.13 (0.96) | 8.12 (0.92)
Baseline Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Population: The analysis population included all randomized participants who have received at least one dose of investigational product and had a baseline FPG measurement.
  mg/dL
    number analyzed (Participants) | 167 | 168 | 166 | 501
    (all) | 170.1 (36.0) | 167.3 (41.1) | 165.8 (37.6) | 167.8 (38.3)
Baseline estimated glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  mL/min/1.73 m^2 | 97.9 (19.2) | 100.2 (19.8) | 99.9 (20.2) | 99.3 (19.7)
Country [Count of Participants; unit: Participants] — Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  Participants
    China | 136 | 135 | 135 | 406
    Hong Kong | 10 | 10 | 7 | 27
    Korea, Republic of | 13 | 10 | 9 | 32
    Philippines | 7 | 8 | 8 | 23
    Taiwan | 4 | 6 | 8 | 18
Anti-hyperglycemic Agent (AHA) Status at Screening (Metformin Alone OR Metformin + Another AHA) [Count of Participants; unit: Participants] — Background AHA therapy at screening. Combination blood glucose lowering agents were counted twice, under each component of the combination. Population: The analysis population included all randomized participants who received at least one dose of investigational product.
  Participants
    Metformin alone | 111 | 121 | 121 | 353
    Metformin + Another AHA | 59 | 48 | 46 | 153
Gender (China Substudy) [Count of Participants; unit: Participants] — Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
  Participants
    number analyzed (Participants) | 136 | 135 | 135 | 406
    Female | 65 | 51 | 66 | 182
    Male | 71 | 84 | 69 | 224
Age Continuous (China Substudy) [Mean (Standard Deviation); unit: Years] — Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
  Years
    number analyzed (Participants) | 136 | 135 | 135 | 406
    (all) | 56.0 (9.0) | 56.2 (9.4) | 56.8 (8.6) | 56.3 (9.0)
Body Weight (China Substudy) [Mean (Standard Deviation); unit: Kilograms] — Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
  Kilograms
    number analyzed (Participants) | 136 | 135 | 135 | 406
    (all) | 71.4 (11.1) | 70.2 (10.2) | 70.6 (12.2) | 70.7 (11.2)
Baseline A1C (China Substudy) [Mean (Standard Deviation); unit: Percentage A1C] — A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and had a baseline A1C measurement.
  Percentage A1C
    number analyzed (Participants) | 135 | 135 | 134 | 404
    (all) | 8.22 (0.94) | 8.13 (0.96) | 8.09 (0.98) | 8.14 (0.96)
Baseline FPG (China Substudy) [Mean (Standard Deviation); unit: mg/dL] — Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and had a baseline FPG measurement.
  mg/dL
    number analyzed (Participants) | 135 | 134 | 134 | 403
    (all) | 175.7 (36.2) | 170.5 (43.0) | 165.5 (37.9) | 170.6 (39.3)
Baseline eGFR (China Substudy) [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
  mL/min/1.73 m^2
    number analyzed (Participants) | 136 | 135 | 135 | 406
    (all) | 99.8 (19.0) | 102.7 (19.8) | 100.8 (21.1) | 101.1 (19.9)
Anti-AHA status at Screening (Metformin Alone OR Metformin + Another AHA) (China Substudy) [Count of Participants; unit: Participants] — Background AHA therapy at screening. Combination blood glucose lowering agents were counted twice, under each component of the combination. Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
  Participants
    Metformin Alone: number analyzed (Participants) | 136 | 135 | 135 | 406
    Metformin Alone | 85 | 92 | 93 | 270
    Metformin + Another AHA: number analyzed (Participants) | 136 | 135 | 135 | 406
    Metformin + Another AHA | 51 | 43 | 42 | 136

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C (%) at Week 26 (Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 26 A1C minus the Week 0 A1C (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants who received at least one dose of investigational product and who had at least one assessment of the respective endpoint at baseline or post baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage A1C
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage A1C | -1.00 [-1.12 to -0.88] | -0.89 [-1.01 to -0.77] | -0.20 [-0.33 to -0.08]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; The primary hypothesis of the study was the mean change from baseline in HbA1c for 15 mg ertugliflozin is greater than that for placebo; Test type: Superiority — Constrained longitudinal data analysis (cLDA); p < 0.001, cLDA — cLDA model with fixed effects for treatment, time, anti-AHA status at Screening (metformin alone, metformin + another AHA), country (China, other), baseline eGFR (continuous) and the interaction of time by treatment; Least squares means = LSM; Difference in the LSM vs. placebo = -0.69, 95% CI 2-sided [-0.85 to -0.52]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; The primary hypothesis of the study was the mean change from baseline in HbA1c for 5 mg ertugliflozin is greater than that for placebo; Test type: Superiority — cLDA model with fixed effects for treatment, time, anti-AHA status at Screening (metformin alone, metformin + another AHA), country (China, other), baseline eGFR (continuous) and the interaction of time by treatment; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -0.80, 95% CI 2-sided [-0.97 to -0.63]

2. Primary Outcome: Change From Baseline in A1C (%) at Week 26 (Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 1
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and who had at least one assessment of the respective endpoint at baseline or post baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage A1C
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage A1C | -1.01 [-1.14 to -0.87] | -0.92 [-1.05 to -0.79] | -0.24 [-0.38 to -0.10]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority; p < 0.001, cLDA — cLDA model with fixed effects for treatment, time, anti-AHA status at Screening (metformin alone, metformin + another AHA), baseline eGFR (continuous) and the interaction of time by treatment; Difference in the LSM vs. placebo = -0.68, 95% CI 2-sided [-0.86 to -0.50]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — cLDA model with fixed effects for treatment, time, anti-AHA status at Screening (metformin alone, metformin + another AHA), baseline eGFR (continuous) and the interaction of time by treatment; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -0.76, 95% CI 2-sided [-0.95 to -0.58]

3. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE) (Including Rescue Approach)
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 28 weeks
Population: The analysis population included all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage of participants | 56.5 | 53.3 | 59.3
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Other; Difference in % vs. Placebo = -6.0, 95% CI 2-sided [-16.5 to 4.6]; Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Other; Difference in % vs. Placebo = -2.8, 95% CI 2-sided [-13.3 to 7.7]; Miettinen-Nurminen method

4. Primary Outcome: Percentage of Participants Experiencing An Adverse Event (AE) (Including Rescue Approach) (China Subpopulation)
Description: as for outcome 3
Time Frame: Up to 28 weeks
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product .
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage of participants | 54.4 | 50.4 | 59.3
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Other; Difference in % vs. Placebo = -8.9, 95% CI 2-sided [-20.5 to 3.0]; Miettinen-Nurminen method
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Other; Difference in % vs. Placebo = -4.8, 95% CI 2-sided [-16.5 to 6.9]; Miettinen-Nurminen method

5. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE (Including Rescue Approach)
Description: as for outcome 3
Time Frame: Up to 26 weeks
Population: The analysis population included all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage of Participants | 1.2 | 0.6 | 1.8

6. Primary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE (Including Rescue Approach) (China Subpopulation)
Description: as for outcome 3
Time Frame: Up to 26 weeks
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage of Participants | 0.7 | 0.7 | 2.2

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 26 (Excluding Rescue Approach)
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 26 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 26 minus FPG at Week 0) which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants who received at least one dose of investigational product and who had at least one assessment of the respective endpoint at baseline or post-baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
mg/dL | -37.09 [-41.73 to -32.45] | -34.47 [-39.15 to -29.79] | -6.69 [-11.57 to -1.82]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — cLDA model with fixed effects for treatment, time, anti-hyperglycemic medication status at Screening (metformin alone, metformin + another AHA), Country (China, other), baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -27.78, 95% CI 2-sided [-33.85 to -21.70]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -30.40, 95% CI 2-sided [-36.45 to -24.35]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 26 (Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 7
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and who had at least one assessment of the respective endpoint at baseline or post-baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
mg/dL | -39.01 [-43.87 to -34.15] | -36.67 [-41.64 to -31.71] | -10.46 [-15.61 to -5.31]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — cLDA model with fixed effects for treatment, time, anti-hyperglycemic medication status at Screening (metformin alone, metformin + another AHA), baseline eGFR (continuous) and the interaction of time by treatment. Time was treated as a categorical variable; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -26.21, 95% CI 2-sided [-32.41 to -20.01]
Statistical Analysis 2: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -28.55, 95% CI 2-sided [-34.67 to -22.43]

9. Secondary Outcome: Change From Baseline in Body Weight at Week 26 (Excluding Rescue Approach)
Description: The change in body weight from baseline reflects the Week 26 body weight minus the Week 0 body weight (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: The analysis population included all randomized participants and who received at least one dose of investigational product and who had at least one assessment of the respective endpoint at baseline or post-baseline up to Week 26.
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Kilograms | -2.95 [-3.29 to -2.60] | -3.18 [-3.52 to -2.83] | -1.17 [-1.54 to -0.81]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -2.00, 95% CI 2-sided [-2.51 to -1.50]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -1.78, 95% CI 2-sided [-2.28 to -1.28]

10. Secondary Outcome: Change From Baseline in Body Weight at Week 26 (Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 9
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Kilograms
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Kilograms | -3.11 [-3.50 to -2.72] | -3.38 [-3.78 to -2.98] | -1.33 [-1.75 to -0.91]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, cLDA; Difference in LS Means vs. Placebo = -2.05, 95% CI 2-sided [-2.63 to -1.21]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -1.79, 95% CI 2-sided [-2.36 to -1.21]

11. Secondary Outcome: Percentage of Participants With HbA1c of <7.0% (53 mmol/Mol) (Logistic Regression Using Multiple Imputation Based on cLDA Model: Excluding Rescue Approach)
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage of participants | 38.2 | 40.8 | 16.2
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — Adjusted odds ratio based on a logistic regression model fitted with fixed effects for treatment anti-hyperglycemic medication status at screening (metformin alone, metformin + another AHA), Country (China, other), baseline eGFR (continuous) and baseline A1C (continuous). Missing data imputed using the cLDA model fitted with fixed effects as in the primary analysis; p < 0.001, Logistic regression model; Adjusted Odds Ratio relative to placebo = 4.56, 95% CI 2-sided [2.49 to 8.35]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p < 0.001, Logistic regression model; Adjusted Odds Ratio relative to placebo = 4.59, 95% CI 2-sided [2.52 to 8.36]

12. Secondary Outcome: Percentage of Participants With HbA1c of <7.0% (53 mmol/Mol) (Logistic Regression Using Multiple Imputation Based on cLDA Model: Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 11
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage of participants | 35.3 | 42.2 | 18.5
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — Adjusted odds ratio based on a logistic regression model fitted with fixed effects for treatment anti-hyperglycemic medication status at screening (metformin alone, metformin + another AHA), baseline eGFR (continuous) and baseline A1C (continuous). Missing data imputed using the cLDA model fitted with fixed effects as in the primary analysis; p < 0.001, Logistic regression model; Adjusted Odds Ratio relative to placebo = 4.49, 95% CI 2-sided [2.32 to 8.68]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 12, analysis 1]; p < 0.001, Logistic regression model; Adjusted Odds Ratio relative to placebo = 3.47, 95% CI 2-sided [1.77 to 6.80]

13. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 26 sitting systolic blood pressure (SBP) minus the Week 0 sitting SBP (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
mmHg | -5.09 [-6.78 to -3.40] | -3.87 [-5.58 to -2.16] | 0.22 [-1.58 to 2.01]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -4.09, 95% CI 2-sided [-6.48 to -1.69]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p < 0.001, cLDA; Difference in the LS Means vs. Placebo = -5.30, 95% CI 2-sided [-7.68 to -2.92]

14. Secondary Outcome: Change From Baseline in Sitting Systolic Blood Pressure at Week 26 (Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 13
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
mmHg | -5.64 [-7.53 to -3.75] | -4.19 [-6.14 to -2.25] | -1.56 [-3.61 to 0.49]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.058, cLDA; Difference in the LS Means vs. Placebo = -2.64, 95% CI 2-sided [-5.36 to 0.09]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.003, cLDA; Difference in the LS Means vs. Placebo = -4.08, 95% CI 2-sided [-6.78 to -1.39]

15. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 26 (Excluding Rescue Approach)
Description: This change from baseline reflects the Week 26 sitting diastolic blood pressure (DBP) minus the Week 0 sitting DBP (which is estimated on average for each treatment group using a constrained longitudinal data analysis model, which allows for participants with missing data to be included in the analysis). Participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment. Per protocol, this data set excludes data for any participant after the initiation of glycemic rescue therapy.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
mmHg | -2.38 [-3.51 to -1.25] | -2.36 [-3.50 to -1.22] | -0.96 [-2.16 to 0.24]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.086, cLDA; Difference in the LS Means vs. Placebo = -1.40, 95% CI 2-sided [-3.00 to 0.20]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 7, analysis 1]; p = 0.081, cLDA; Difference in the LS Means vs. Placebo = -1.42, 95% CI 2-sided [-3.01 to 0.17]

16. Secondary Outcome: Change From Baseline in Sitting Diastolic Blood Pressure at Week 26 (Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 15
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
mmHg | -2.82 [-4.11 to -1.54] | -2.77 [-4.09 to -1.45] | -1.82 [-3.21 to -0.43]
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.315, cLDA; Difference in the LS Means vs. Placebo = -0.95, 95% CI 2-sided [-2.80 to 0.90]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Superiority — [test comment as in outcome 8, analysis 1]; p = 0.282, cLDA; Difference in the LS Means vs. Placebo = -1.00, 95% CI 2-sided [-2.83 to 0.83]

17. Secondary Outcome: Percentage of Participants With HbA1c of <6.5% (48 mmol/Mol) at Week 26 (Logistic Regression Using Multiple Imputation: Excluding Rescue Approach)
Description: as for outcome 11
Time Frame: Week 26
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage of participants | 14.7 | 15.4 | 2.4
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p = 0.001, Logistic regression model — Nominal p-values were provided; Adjusted Odds Ratio relative to placebo = 8.90, 95% CI 2-sided [2.46 to 32.22]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p < 0.001, Logistic regression model — Nominal p-values were provided; Adjusted Odds Ratio relative to placebo = 10.69, 95% CI 2-sided [2.95 to 38.71]

18. Secondary Outcome: Percentage of Participants With HbA1c of <6.5% (48 mmol/Mol) at Week 26 (Logistic Regression Using Multiple Imputation: Excluding Rescue Approach) (China Subpopulation)
Description: as for outcome 11
Time Frame: Week 26
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage of participants | 14.7 | 17.0 | 3.0
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Superiority — [test comment as in outcome 11, analysis 1]; p < 0.001, Logistic regression model — Nominal p-values were provided; Adjusted Odds Ratio relative to placebo = 8.34, 95% CI 2-sided [2.52 to 27.60]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg; Test type: Superiority — Adjusted odds ratio based on a logistic regression model fitted with fixed effects for treatment, anti-hyperglycemic medication status at screening (metformin alone, metformin + another AHA), baseline eGFR (continuous) and baseline A1C (continuous). Missing data imputed using the cLDA model fitted with fixed effects as in the primary analysis; p < 0.001, Logistic regression model — Nominal p-values were provided; Adjusted Odds Ratio relative to placebo = 8.29, 95% CI 2-sided [2.44 to 28.11]

19. Secondary Outcome: Percentage of Participants Requiring Glycemic Rescue Therapy Through Week 26.
Description: Per protocol, participants who met pre-specified glycemic criteria were rescued with oral tablets of open-label glimepiride and dosed according to Investigator judgment.
Time Frame: Week 26
Population: The analysis population included all randomized participants who received at least one dose of investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 167
Percentage of Participants | 1.2 | 0.6 | 9.6
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen method; Miettinen & Nurminen method stratified by country ('China' or 'other') for the overall population; Difference in % (Ert. 15 mg. - placebo) = -9.0, 95% CI [-14.5 to -5.0]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen method; Miettinen & Nurminen method stratified by country ('China' or 'other') for the overall population; Difference in % (Ert. 5 mg. - placebo) = -8.4, 95% CI 2-sided [-14.0 to -4.4]

20. Secondary Outcome: Percentage of Participants Requiring Glycemic Rescue Therapy Through Week 26 (China Subpopulation)
Description: as for outcome 19
Time Frame: Week 26
Population: as for outcome 6
Measure: Number; unit: Percentage of Participants
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 135
Percentage of Participants | 0.0 | 0.7 | 9.6
Statistical Analysis 1: Comparison: Ertugliflozin 15 mg vs Placebo; Test type: Other; p = 0.001, Miettinen & Nurminen method; Difference in % (Ert. 15 mg. - placebo) = -8.9, 95% CI [-15.1 to -4.2]
Statistical Analysis 2: Comparison: Ertugliflozin 5 mg vs Placebo; Test type: Other; p < 0.001, Miettinen & Nurminen method; Difference in % (Ert. 5 mg. - placebo) = -9.6, 95% CI 2-sided [-15.8 to -5.7]

21. Secondary Outcome: Time to Glycemic Rescue Therapy
Description: as for outcome 19
Time Frame: Up to 183 days
Population: The analysis population included all randomized participants who received at least one dose of investigational product who received glycemic rescue through Week 26.
Measure: Median (Full Range); unit: Days
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 2 | 1 | 16
Days | NA [41 to 85] — The median is not estimable due to the low number of participants rescued. | NA [149 to 149] — The median is not estimable due to the low number of participants rescued. | NA [22 to 183] — The median is not estimable due to the low number of participants rescued.

22. Secondary Outcome: Time to Glycemic Rescue Therapy (China Subpopulation)
Description: as for outcome 19
Time Frame: Up to 149 days
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and who received glycemic rescue through Week 26. No participants in the Ertugliflozin 5 mg group were rescued.
Measure: Median (Full Range); unit: Days
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 0 | 1 | 13
Days |  | NA [149 to 149] — The median is not estimable due to the low number of participants rescued. | NA [22 to 145] — The median is not estimable due to the low number of participants rescued.

23. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: No ertugliflozin plasma concentrations were determined for participants receiving placebo. Lower limit of quantification for ertugliflozin was 0.500 ng/mL.
Time Frame: Week 6: Pre-Dose
Population: The analysis population included all randomized participants who received at least one dose of investigational product and who had at least one plasma concentration value above the lower limit of quantification. No ertugliflozin plasma concentrations were determined for participants receiving placebo.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 9.17 (18.39) | 24.59 (43.84) |

24. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: as for outcome 23
Time Frame: Week 12: Pre-Dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 8.18 (15.25) | 27.11 (66.02) |

25. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: as for outcome 23
Time Frame: Week 12: 60 min. Post-Dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 91.49 (50.61) | 277.60 (130.66) |

26. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: as for outcome 23
Time Frame: Week 18: Pre-Dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 6.59 (12.53) | 17.54 (24.62) |

27. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: as for outcome 23
Time Frame: Week 18: 60 min. Post-Dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 91.40 (44.77) | 274.23 (146.14) |

28. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach
Description: as for outcome 23
Time Frame: Week 26: Pre-Dose
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 170 | 169 | 0
ng/mL | 7.34 (14.18) | 26.66 (62.17) |

29. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 6: Pre-Dose
Population: The analysis population included all randomized participants in China who received at least one dose of investigational product and who had at least one plasma concentration value above the lower limit of quantification. No ertugliflozin plasma concentrations were determined for participants receiving placebo.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 0
ng/mL | 7.88 (14.88) | 22.29 (42.81) |

30. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 12: Pre-Dose
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 136 | 135 | 0
ng/mL | 7.40 (12.21) | 23.84 (52.64) |

31. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 12: 60 min. Post-Dose
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 131 | 125 | 0
ng/mL | 97.36 (48.98) | 294.49 (124.73) |

32. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 18: Pre-Dose
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 127 | 125 | 0
ng/mL | 6.30 (11.50) | 17.07 (27.06) |

33. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 18: 60 min. Post-Dose
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 127 | 125 | 0
ng/mL | 94.82 (41.40) | 285.28 (141.59) |

34. Secondary Outcome: Ertugliflozin Plasma Concentrations Summary Statistics Over Time: Including Rescue Approach (China Subpopulation)
Description: as for outcome 23
Time Frame: Week 26: Pre-Dose
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
Number analyzed (Participants) | 127 | 118 | 0
ng/mL | 7.26 (14.09) | 24.91 (57.95) |

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: The analysis population included all randomized and treated participants.
Arm/Group | Ertugliflozin 5 mg | Ertugliflozin 15 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/169 | 0/167
Serious Adverse Events (participants affected / at risk) | 9/170 | 10/169 | 2/167
Other Adverse Events (participants affected / at risk) | 22/170 | 31/169 | 44/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=170) | Ertugliflozin 15 mg (N=169) | Placebo (N=167)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ertugliflozin 5 mg (N=170) | Ertugliflozin 15 mg (N=169) | Placebo (N=167)
Nasopharyngitis (Infections and infestations) | 9 (13) | 9 (11) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 9 (9) | 14 (16)
Hyperuricaemia (Metabolism and nutrition disorders) | 5 (5) | 9 (9) | 20 (21)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (10) | 9 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to the sponsor at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT02630706/Prot_SAP_000.pdf